CLINICAL TRIAL: NCT05558800
Title: Bone-To-Implant Contact At 4- And 6-Week Healing Stages in Implants Having Either Machined, SLA Medium Roughness, Nanostructured Calcium-Incorporated or Plasma Reactivated Nanostructured Calcium-Incorporated Surface: A Histologic Study.
Brief Title: Bone-To-Implant Contact At 4- And 6-Week Healing Stages in Implants With Different Surfaces.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Christian Makari, Associate Professor, Saint-Joseph University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: XFMD171
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Implant Geometry

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Xpeed (Active Comparator): Implant with Xpeed surface
  Interventions: Procedure: Implant placement
- SLA surface (Active Comparator): Implant with SLA surface
  Interventions: Procedure: Implant placement
- Machined (Placebo Comparator): Implant with machined surface
  Interventions: Procedure: Implant placement
- XPEEDActive (Active Comparator): Implant with plasma treatment reactivated XPEED implant surface
  Interventions: Procedure: Implant placement

INTERVENTIONS:
Procedure: Implant placement — Implant placement with different surface types

SUMMARY:
Objective: Implant surface topography is a key element in achieving osseointegration. Nanostructured surfaces have shown promising results in accelerating and improving bone healing around dental implants. The main objective of the present clinical study is to compare, at 4 and 6w, bone-to-implant contact in implants having either machined surface (MAC), SLA medium roughness surface or a Nanostructured Calcium-Incorporated surface (XPEED®). Thirty five mini-implants with 3 different surface treatments (XPEED® (n=16) - SLA (n=13) - Machined (n=6)), were placed in the posterior maxilla of 11 patients then retrieved at either 4 or 6w in a randomized split-mouth study design.

ELIGIBILITY:
Inclusion Criteria:

* • Height of the residual bone crest in the programmed implant site ≥ 9 mm and thickness ≥ 7mm.

  * Availability, in each sector, of sufficient mesio-distal space allowing placement of 2 standard-sized implants and at least 2 mini-implants (3.5x8.5mm) for retrieval.
  * Healed bone crest (≥ 3 months elapsed after extraction or tooth loss).
  * Age > 18 years.
  * Ability to examine and fully understand the study protocol.

Exclusion Criteria:

* • Myocardial infarction within the past 6 months.

  * Poorly controlled diabetes (HBA1c > 7.5%).
  * Coagulation disorders.
  * Radiotherapy to the head/neck area within the past two years.
  * Present or past treatment with intravenous bisphosphonates.
  * Immunocompromised patients.
  * Psychological or psychiatric problems.
  * Alcohol or drug abuse.
  * Poor oral hygiene and motivation (full mouth plaque score > 30% and/or full mouth bleeding score > 20%).
  * Uncontrolled periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Bone to implant contact | 4 weeks healing period after implant placement
  Histology technique on specimen retrieved containing mini-implants and bone surrounding it
Bone to implant contact | 6 weeks healing period after implant placement
  Histology technique on specimen retrieved containing mini-implants and bone surrounding it

CONTACTS AND LOCATIONS:
Overall Officials: Christian Makary, Phd, Principal Investigator — Saint Joseph University - Beirut
Locations (1):
- Saint Joseph University, Beirut, Lebanon